CLINICAL TRIAL: NCT01764373
Title: Pilot Study of Exercise and Peripheral Nerve Function in People With Diabetes - Exercise and Neuropathy Research Group v.2 (ENRGy2) Addendum
Brief Title: Pilot Study of Exercise and Peripheral Nerve Function in People With Diabetes - ENRGy2 Addendum
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Kansas (Other)
Responsible Party: Principal Investigator, Patricia Kluding, PhD, Associate Professor, University of Kansas
Organization: University of Kansas Medical Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: ENRGy2 Addendum
Record Dates: First submitted 2013-01-07; First posted 2013-01-09 (Estimated); Last update posted 2013-09-27 (Estimated); Status verified 2013-09

CONDITIONS: Diabetic Neuropathy
Keywords: Pain; Fitness; Diabetes; Aerobic Exercise
MeSH Terms: conditions — Diabetic Neuropathies; Pain; Diabetes Mellitus | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 16-Week Exercise Program (Experimental): Subjects to participate in 16-week3 supervised aerobic exercise 3 times per week. Exercise sessions to last between 30 and 60 minutes.
  Interventions: Other: Aerobic Exercise

INTERVENTIONS:
Other: Aerobic Exercise — Aerobic exercises in the program include cycle ergometers, treadmills, recumbent steppers and elliptical trainers.

SUMMARY:
This is an amendment to study posting NCT00970060. Based on preliminary results from that study is was determined there needs to be a follow-up exercise intervention study. This study has two additional aims than the original study. The objectives are to determine is a prolonged exercise routine, 16-weeks, paired with refined measures of effectiveness positively impact people with diabetic neuropathy.

ELIGIBILITY:
Inclusion Criteria:

* Age 40-70
* Type 2 diabetes
* Peripheral neuropathy

Exclusion Criteria:

* serious cardiac pathology such as recent myocardial infarction or heart surgery, uncontrolled cardiac arryhthmia, hypertrophic cardiomyopathy symptomatic aortic stenosis or heart failure, unstable angina, acute pulmonary embolus or myocarditis, conduction abnormalities, or mitral valve prolapse
* serious musculoskeletal problems that would limit ability to exercise
* skin conditions, circulatory insufficiency, or open wounds in the leg that would interfere with healing from the biopsy
* open wounds on the weight bearing surface of the feet
* not able to ambulate independently
* stroke or other central nervous system pathology
* stage 2 hypertension (resting blood pressure > 160 systolic or > 100 diastolic)
* lidocaine allergy
* anticipated difficulty with blood clotting due to Coumadin(Warfarin) use or blood clotting disorder
* body weight > 450 lbs
* inadequate cognition and communication abilities, defined as < 24 on the Mini Mental Status Exam (MMSE)
* pregnant or planning on becoming pregnant in the 18 weeks following enrollment

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2012-06; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Change nerve function | Baseline to Week 16
  Change in nerve function will be quantified using the Total Neuropathy Score (TNS). The TNS is a composite measure of peripheral nerve function that includes grading of signs/symptoms, nerve conduction studies, and quantitative sensory testing. We will not include proprioceptive testing in this project.
Change in aerobic fitness | Baseline to Week 16
  Aerobic fitness will be assessed with a graded maximal exercise test as in the previous protocol with a metabolic cart and integrated ECG.

SECONDARY OUTCOMES:
Change in cutaneous innervation | Baseline to Week 16
  Change will be measured after exercise intervention to see what effects exercise has on dermal and epidermal innervation. Change measured via skin biopsy.
Change in maximal workload | Baseline to Week 16
  Measured as part of the aerobic fitness assessment. Use of standardized protocol with total body recumbent stepped to be used to obtain the maximal workload.
Change in pain experienced | Baseline to Week 16
  Pain will be measured using the Brief Pain Inventory Short Form for diabetic peripheral neuropathy. This scale has been specifically validated in this population and consists of 3 pain severity items and a 7-item pain interference scale.

CONTACTS AND LOCATIONS:
Overall Officials: Patricia Kluding, PhD, Principal Investigator — University of Kansas Medical Center
Locations (1):
- University of Kansas Medical Center, Kansas City, Kansas, United States

REFERENCES:
- [Derived] Kluding PM, Pasnoor M, Singh R, D'Silva LJ, Yoo M, Billinger SA, LeMaster JW, Dimachkie MM, Herbelin L, Wright DE. Safety of aerobic exercise in people with diabetic peripheral neuropathy: single-group clinical trial. Phys Ther. 2015 Feb;95(2):223-34. doi: 10.2522/ptj.20140108. Epub 2014 Oct 2. PMID 25278335
- See also: Original Protocol Study Posting — http://clinicaltrials.gov/ct2/show/NCT00970060